CLINICAL TRIAL: NCT02863302
Title: Reflexology Treatment for Newly Diagnosed AML Patients, Can it Reduce GI Tract Side Effects, and Improve and Improve Patients Mood.
Brief Title: Reflexology: An Intervention for Acute Myeloid Leukemia(AML) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Netanel Horowitz MD, Head of ambulatory unit , hematology division, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0107-16
Record Dates: First submitted 2016-07-10; First posted 2016-08-11 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia, Reflexology
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reflexology treatment (Experimental): All patients will receive reflexology (a specialized foot therapy) from a certified reflexologist twice weekly from the beginning of chemotherapy treatment until the end of hospitalization.
  Interventions: Other: Reflexology treatment

INTERVENTIONS:
Other: Reflexology treatment — All patients will receive reflexology (a specialized foot therapy) from a certified reflexologist twice weekly from the beginning of chemotherapy treatment.

SUMMARY:
The aim of this study is to test a complementary therapy intervention (reflexology) that will assist in improving quality of life (QOL) for patients undergoing chemotherapy for acute myeloid leukemia. within the context of conventional medical care. Quality of life will be assessed via intermediate indicators: 1) physical indicators (greater physical functioning, lower presence of symptoms) 2) emotional indicators (greater spirituality, lower anxiety, and lower depressive symptomology); by a specific questionnaire. 3) chemotherapy side effects associated with the digestive system.

DETAILED DESCRIPTION:
The goal of this study is to test a complementary therapy intervention that will assist in improving quality of life (QOL) for patients undergoing chemotherapy for acute myeloid leukemia within the context of conventional medical care. This open study will test a one group design in which participants will continue to receive conventional care. All patients will receive reflexology (a specialized foot therapy) from a certified reflexologist twice weekly from the beginning of chemotherapy treatment.

The specific aims are: 1) to evaluate the effect of reflexology treatment on chemotherapy side effects effecting the digestive system. 2) to evaluate the effect of reflexology treatment on Quality of life. The assessment of the treatment will be executed on the FACIT-D VERSION 3.The influences of the treatment will also be evaluated by the nursing staff, in order to describe the patient's mental health and the condition of his intestinal movement.The side effect before during and after the chemotherapy treatment will be compared using the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of AML
* chemotherapy treatment
* signing a consent form.

Exclusion Criteria:

• Not willing to sign a consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the FACIT-D questionaire. | Change from baseline in the FACIT-D questionaire at 1,2,3, and 4 weeks from the beginning of chemotherapy treatment.

SECONDARY OUTCOMES:
To evaluate the effect of reflexology treatment on chemotherapy associated diarrhea | Diarrhea frequency will be recorded daily from the first day of chemotherapy and up to 30 days.
  Diarrhea frequency will be recorded daily by the nursing staff and entered into the patients medical chart.

CONTACTS AND LOCATIONS:
Overall Officials: Netanel A Horowitz, MD, Principal Investigator — Rambam Health Care Campus, Haifa, Israel.
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rahbar MH, Wyatt G, Sikorskii A, Victorson D, Ardjomand-Hessabi M. Coordination and management of multisite complementary and alternative medicine (CAM) therapies: experience from a multisite reflexology intervention trial. Contemp Clin Trials. 2011 Sep;32(5):620-9. doi: 10.1016/j.cct.2011.05.015. Epub 2011 Jun 2. PMID 21664296
- [Result] Sikorskii A, Wyatt G, Victorson D, Faulkner G, Rahbar MH. Methodological issues in trials of complementary and alternative medicine interventions. Nurs Res. 2009 Nov-Dec;58(6):444-51. doi: 10.1097/NNR.0b013e3181bf15fe. PMID 19918155